CLINICAL TRIAL: NCT06092905
Title: Endoscopic Common Bile Duct Stones Clearance During Pregnancy: Challenges and Solutions
Brief Title: Endoscopic Common Bile Duct Stones Clearance During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Abdallah Mohamed Taha Aly, Assistant Professor, South Valley University
Other Study IDs: SVU-MED-SUR11-4-23-3-601
Record Dates: First submitted 2023-10-15; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Common Bile Duct Calculi
Keywords: Common Bile Duct Stones; Endoscopic clearance; Jaundice; Pregnancy
MeSH Terms: conditions — Gallstones; Jaundice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with symptomatic common bile duct stones: Pregnant women with symptomatic common bile duct stones
  Interventions: Other: Endoscopic clearance of common bile duct stones

INTERVENTIONS:
Other: Endoscopic clearance of common bile duct stones — Under general anesthesia, in left lateral decubitus, endoscopic clearance of common bile duct stones was done. Ultrasonography was used to ensure right positioning of the guide wire in the common bile duct, and ensure stone clearance.

SUMMARY:
Background: Pregnancy is associated with a higher risk of common bile duct stones. Currently Endoscopic Retrograde Cholangiopancreatography (ERCP) is the treatment of choice for symptomatic choledocholithiasis. However, ERCP during pregnancy is associated with hazards of radiation exposure, as well as challenging patient positioning and anesthesia

DETAILED DESCRIPTION:
This is a retrospective analysis of endoscopic common bile duct stone clearance in pregnant patients with symptomatic choledocholithiasis between June 2015 and June 2023.

Sedation and anesthesia was done by safe medications by senior anesthetist, and the endoscopic procedure was performed in left lateral decubitus instead of prone position. The gravid uterus was kept away from the monopolar electrocautery current pathway. Radiocontrast injection and fluoroscopy was deleted and replaced by trans-abdominal US and endoscopic bile aspiration Data including perioperative outcomes and follow up data will collected, tabulated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with symptomatic common bile duct stones.

Exclusion Criteria:

* Presence of pancreatitis or cholangitis.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant woman with symptomatic common bile duct stones
Study Population: Pregnant women, presented with symptomatic common bile duct stones to the general surgery department at Qena University Hospital, South Valley University, Egypt, between June 2015 and June 2023. Endoscopy was performed for clearance of the stones.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Complications | Till one month after delivery.
  any perioperative complications as pancreatitis, perforation, bleeding, abortion, preterm labor.

CONTACTS AND LOCATIONS:
Overall Officials: ABDALLAH M ALY, MD, Principal Investigator — South Valley University
Locations (1):
- Qena Faculty of Medicine, South Valley University Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luo L, Zen H, Xu H, Zhu Y, Liu P, Xia L, He W, Lv N. Clinical characteristics of acute pancreatitis in pregnancy: experience based on 121 cases. Arch Gynecol Obstet. 2018 Feb;297(2):333-339. doi: 10.1007/s00404-017-4558-7. Epub 2017 Nov 21. PMID 29164335
- [Background] Xu Q, Wang S, Zhang Z. A 23-year, single-center, retrospective analysis of 36 cases of acute pancreatitis in pregnancy. Int J Gynaecol Obstet. 2015 Aug;130(2):123-6. doi: 10.1016/j.ijgo.2015.02.034. Epub 2015 May 2. PMID 25983209
- [Background] Goldschmiedt M, Wolf L, Shires T. Treatment of symptomatic choledocholithiasis during pregnancy. Gastrointest Endosc. 1993 Nov-Dec;39(6):812-4. doi: 10.1016/s0016-5107(93)70272-2. No abstract available. PMID 8293907
- [Background] Tham TC, Vandervoort J, Wong RC, Montes H, Roston AD, Slivka A, Ferrari AP, Lichtenstein DR, Van Dam J, Nawfel RD, Soetikno R, Carr-Locke DL. Safety of ERCP during pregnancy. Am J Gastroenterol. 2003 Feb;98(2):308-11. doi: 10.1111/j.1572-0241.2003.07261.x. PMID 12591046
- [Background] Inamdar S, Berzin TM, Sejpal DV, Pleskow DK, Chuttani R, Sawhney MS, Trindade AJ. Pregnancy is a Risk Factor for Pancreatitis After Endoscopic Retrograde Cholangiopancreatography in a National Cohort Study. Clin Gastroenterol Hepatol. 2016 Jan;14(1):107-14. doi: 10.1016/j.cgh.2015.04.175. Epub 2015 May 5. PMID 25952311